CLINICAL TRIAL: NCT02067975
Title: Neuroimaging of Tryptophan Challenge in People With Schizophrenia and Healthy Controls
Brief Title: Tryptophan MRI in People With Schizophrenia and Healthy Controls
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Tanabe Pharma Corporation (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert Buchanan, Director, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00057861; 1P50MH103222-01 (NIH)
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Results first posted 2021-08-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia
Keywords: tryptophan; kynurenic acid; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Tryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Controls (Other): All participants will receive both 6gm of tryptophan at least two weeks apart at time zero of 7 hour visits 2 and 3, and will also receive Placebo will be a liquid drink without tryptophan. 6mg at least two weeks apart at time zero of the 7 hour visits 2 and 3. The order in which participants receive either placebo or tryptophan will be randomized (ie. placebo first study visit day tryptophan on second study day, or tryptophan on first study day and placebo on second study day)
  Interventions: Drug: Tryptophan; Drug: Placebo
- Schizophrenia Related Disorders (Other): All participants will receive both 6gm of tryptophan at least two weeks apart at time zero of 7 hour visits 2 and 3, and will also receive Placebo will be a liquid drink without tryptophan. 6mg at least two weeks apart at time zero of the 7 hour visits 2 and 3. The order in which participants receive either placebo or tryptophan will be randomized (ie. placebo first study visit day tryptophan on second study day, or tryptophan on first study day and placebo on second study day)
  Interventions: Drug: Tryptophan; Drug: Placebo

INTERVENTIONS:
Drug: Tryptophan
Drug: Placebo

SUMMARY:
Kynurenic acid (KYNA) is a naturally occurring chemical in the brain. Studies with rodents indicate that levels of KYNA can impact levels of the neurotransmitters glutamate and dopamine. One way to reliably increase KYNA levels is by ingesting the amino acid tryptophan. Tryptophan is a normal part of the human diet. Tryptophan gets metabolized/changed to other chemicals in the body- including KYNA. By giving people 6 grams of tryptophan, the investigators will be able to increase the KYNA level in a controlled way. The investigators will then be able to study the effects of KYNA on neurotransmitters by using cognitive tests and magnetic resonance imaging techniques (measuring brain activity and brain chemistry using the MRI magnet). They will test people using tryptophan and also using a placebo to look for differences. The investigators will test healthy controls and people with schizophrenia to look for differences.

DETAILED DESCRIPTION:
There is emerging evidence to suggest that disturbances in the kynurenine pathway may be related to the pathophysiology of schizophrenia. Several post-mortem studies have documented specific abnormalities in the kynurenine pathway, including increased levels of kynurenine and kynurenic acid (KYNA) in the prefrontal cortex of people with schizophrenia (1-4). Increased levels of kynurenine and KYNA have also been observed in the cerebral spinal fluid (CSF) of people with this illness (5). In addition, post-mortem studies have documented changes in key enzymes, including increased expression of tryptophan 2,3-dioxygenase (2, 6) (TDO), which converts tryptophan to kynurenine, and reduced activity of kynurenine 3-monooxygenase (KMO) (4), which may shift metabolism towards enhanced KYNA formation. Finally, a number of genetic studies have implicated the KYNA pathway in this disease. Wonodi et al. (7) found decreased KMO gene expression in the frontal eye field of people with schizophrenia, and Holtze et al. (8) recently reported an association between a KMO SNP and CSF levels of KYNA. Notably, although the exact mechanism underlying the KP impairment in people with schizophrenia is unknown, immune and stress mechanisms have been implicated (7,9).

Increased KYNA may have a number of adverse consequences of importance in schizophrenia. In particular, KYNA is an antagonist of the α7 nicotinic and NMDA glutamate receptors. Dysfunctions of these receptors have been linked to the cognitive impairments and symptom manifestations observed in people with schizophrenia. The purpose of the proposed project is to examine the impact of increased brain KYNA on performance of cognitive tasks and related neuroimaging measures in people with DSM-5/DSM-IV-TR schizophrenia, schizophreniform, or schizoaffective disorder patients and healthy controls. In addition, the investigators will secondarily investigate the relationship of peripheral inflammatory markers and glucocorticoid levels as part of the HPA stress axis to examine relationships and shift to a Type 2 immune response in schizophrenia. Using tryptophan loading to increase KYNA levels, the study will test the hypothesis, based on complementary preliminary studies in rodents, that disease-related cognitive deficits in people with schizophrenia are preferentially susceptible to (further) elevations in KYNA levels.

The investigators hypothesize that tryptophan-induced elevations in brain KYNA levels will: 1) acutely impair performance on measures of verbal and visual memory, attention, working memory, and processing speed in people with schizophrenia; 2) alter dorsolateral-hippocampal activation and connectivity, which underlies the performance of the relational memory task; and 3) decrease mPFC MRS measures of glutamate, consistent with preclinical microdialysis data. In an exploratory framework, the investigators hypothesize that increased brain KYNA levels alter default network activation and connectivity, an effect which may be mediated by the action of KYNA on α7 nicotinic and/or NMDA receptors. The investigators will also investigate the extent to which cytokine and HPA axis peripheral measures are related to the effect of tryptophan-induced elevated KYNA levels on cognitive performance and fMRI and MRS measures. Comparisons with results from healthy controls will determine if participants with schizophrenia have an aberrant or exaggerated response to increased KYNA levels.

Funding Information:

Funded by the National Institute of Mental Health (NIMH)

Grant Number- 1P50MH103222-01

Principal Investigator- Robert Schwarcz, PhD

Project Title- Kynurenic Acid and Cognitive Abnormalities in Schizophrenia

Program Officer Full Name- Steven Zalcamn

External Org# Name- University of Maryland, Baltimore

ELIGIBILITY:
Inclusion Criteria (Schizophrenia:

* Males and females between the ages of 18 and 55 years
* Has met DSM-IV-TR/DSM-5 Criteria for schizophrenia, schizoaffective disorder or schizophreniform disorder
* Prescription of antipsychotic medication for at least 60 days and constant dose for 30 days prior to study entry (either first or second generation antipsychotics permitted)
* Women must be in the first half of their menstrual cycle at the time of the 2 challenge visits

Inclusion Criteria (Healthy Controls):

* Males and females between the ages of 18 and 55 years
* No DSM-IV-TR/DSM-5 Axis I Disorder (documented by SCID)
* Women must be in the first half of their menstrual cycle at the time of the 2 challenge visits

Exclusion Criteria:

* DSM-IV-TR/DSM-5 substance abuse in the last month or substance dependence in the last 6 months (documented by SCID)
* Calgary Depression Scale total score ≥ 10 at baseline
* Current smoker (expired CO ≥ 10 ppm)
* Current use of nicotine replacement therapy or other nicotine products
* Pregnancy or breast feeding
* Post-menopausal women will not be included due to changes in the HPA axis expression and hormonal effects on cognition. In women over the age of 45, menopausal status will be evaluated clinically
* Excessive self-reported daily caffeine intake, defined as intake exceeding 1000 mg or the equivalent of 8 cups of coffee
* Active disorders that have been reported to affect tryptophan metabolism or interfere with absorption will be excluded (Acute Intermittent Porphyria, Celiac Disease, Crohn's Disease, Irritable Bowel Syndrome
* History of an organic brain disorder; mental retardation; or a medical condition, whose pathology or treatment could alter cognition
* Claustrophobia
* Metal in body that will interfere with MR imaging
* Treatment with monoamine oxidase inhibitors, migraine headache medications (triptans) and dextromethorphan

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- [Derived] Hare SM, Adhikari BM, Mo C, Chen S, Wijtenburg SA, Seneviratne C, Kane-Gerard S, Sathyasaikumar KV, Notarangelo FM, Schwarcz R, Kelly DL, Rowland LM, Buchanan RW. Tryptophan challenge in individuals with schizophrenia and healthy controls: acute effects on circulating kynurenine and kynurenic acid, cognition and cerebral blood flow. Neuropsychopharmacology. 2023 Oct;48(11):1594-1601. doi: 10.1038/s41386-023-01587-3. Epub 2023 Apr 28. PMID 37118058

RESULTS

PARTICIPANT FLOW:
Groups:
- Schizophrenia Related Disorders: Tryptophan First, Then Placebo; Schizophrenia Related Disorders: Placebo First, Then Tryptophan: All participants received 6gs of placebo on the 2nd visit, and then received 6gs of tryptophan at the 3rd visit no less than two weeks apart at time zero of 7-hour visits 2 and 3. The order in which participants received either placebo or tryptophan was be randomized. The participant and the study staff did not know the order; only the pharmacist distributing the meds knew. These participants were diagnosed with Schizophrenia, Schizoaffective, or Schizophreniform.
- Healthy Control: Tryptophan First, Then Placebo; Healthy Control: Placebo First, Then Tryptophan: All participants received 6gs of placebo on the 2nd visit, and then received 6gs of tryptophan at the 3rd visit no less than two weeks apart at time zero of 7-hour visits 2 and 3. The order in which participants received either placebo or tryptophan was be randomized. The participant and the study staff did not know the order; only the pharmacist distributing the meds knew. These participants had no psychiatric conditions.
- Schizophrenia Related Disorders: Screening Only/Not Randomized: All participants had not yet completed the screening phase or been randomized. These participants were diagnosed with Schizophrenia, Schizoaffective, or Schizophreniform.
- Healthy Control: Screening Only/Not Randomized: All participants had not yet completed the screening phase or been randomized. These participants had no psychiatric conditions.
Period: Overall Study
Arm/Group | Schizophrenia Related Disorders: Tryptophan First, Then Placebo | Healthy Control: Tryptophan First, Then Placebo | Schizophrenia Related Disorders: Placebo First, Then Tryptophan | Healthy Control: Placebo First, Then Tryptophan | Schizophrenia Related Disorders: Screening Only/Not Randomized | Healthy Control: Screening Only/Not Randomized
Started | 20 | 18 | 21 | 18 | 8 | 8
Completed | 16 | 16 | 19 | 14 | 0 | 0
Not Completed | 4 | 2 | 2 | 4 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls; Schizophrenia Related Disorders: All participants will receive both 6gm of tryptophan at least two weeks apart at time zero of 7 hour visits 2 and 3, and will also receive Placebo will be a liquid drink without tryptophan. 6mg at least two weeks apart at time zero of the 7 hour visits 2 and 3. The order in which participants receive either placebo or tryptophan will be randomized (ie. placebo first study visit day tryptophan on second study day, or tryptophan on first study day and placebo on second study day). Note that some of the participants included only participated in the screening and did not participate in the challenge phase of the study.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Schizophrenia Related Disorders | Total
Number analyzed (Participants) | 44 | 49 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 49 | 93
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.75 (11.70) | 35.97959184 (9.847778506) | 35.39784946 (10.72293335)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 20 | 33 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 26 | 44
  White | 19 | 21 | 40
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 49 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in Verbal Memory Scores From Baseline to 4 Hours Post-Treatment
Description: The following assessment was used to assess the outcome measure: the Hopkins Verbal Learning Test-Revised (HVLT-R). HVLT total scores range from 0 to 36. In order to conduct group comparisons, the HVLT raw total scores are converted to a t-score (range: -10 to 80). The mean t-scores for each condition are below (see outcome measure data table). Higher scores represent better performance. Participants performed the same task before pre- and post-treatment with Tryptophan and again with placebo (2 weeks between conditions). Change in scores pre- and post-treatment were compared between the Tryptophan and placebo conditions.
Time Frame: The order in which participants received either the tryptophan or placebo was randomized. The HVLT was administered 90 minutes prior to treatment and 4 hours post treatment. There were at least two weeks between the challenge days.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthy Controls: Placebo; Schizophrenia Related Disorders: Placebo: All participants received 6gm of placebo dissolved in water. The HVLT was administered 90 minutes prior to placebo and 4 hours post placebo administration.
- Healthy Controls: Tryptophan; Schizophrenia Related Disorders: Tryptophan: All participants received 6gm of tryptophan dissolved in water. The HVLT was administered 90 minutes prior to placebo and 4 hours post placebo administration.
Arm/Group | Healthy Controls: Placebo | Schizophrenia Related Disorders: Placebo | Healthy Controls: Tryptophan | Schizophrenia Related Disorders: Tryptophan
Number analyzed (Participants) | 30 | 37 | 31 | 37
score on a scale | 53.90 (8.01) | 40.49 (11.27) | 53.03 (9.53) | 38.49 (10.77)

ADVERSE EVENTS:
Time Frame: A minimum of 5 weeks (there are a minimum of 2 weeks between visits and there are 3 visits)
Groups:
- Healthy Control: Tryptophan; Schizophrenia Related Disorders: Tryptophan: All participants received 6gm of tryptophan dissolved in water.
- Healthy Controls: Placebo; Schizophrenia Related Disorders: Placebo: All participants received 6gm of placebo dissolved in water.
- Healthy Controls: Screening; Schizophrenia Related Disorders: Screening: All participants had not yet completed the screening phase or been randomized.
Arm/Group | Healthy Control: Tryptophan | Schizophrenia Related Disorders: Tryptophan | Healthy Controls: Placebo | Schizophrenia Related Disorders: Placebo | Healthy Controls: Screening | Schizophrenia Related Disorders: Screening
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/41 | 0/36 | 0/41 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/41 | 0/36 | 0/41 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 13/36 | 6/41 | 0/36 | 3/41 | 1/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control: Tryptophan (N=36) | Schizophrenia Related Disorders: Tryptophan (N=41) | Healthy Controls: Placebo (N=36) | Schizophrenia Related Disorders: Placebo (N=41) | Healthy Controls: Screening (N=8) | Schizophrenia Related Disorders: Screening (N=8)
Nausea (General disorders) | 7 (7) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0) | NA | 1 (1) | 0 (0) | 0 (0)
Vomiting (General disorders) | 4 (4) | 1 (1) | NA | 0 (0) | 0 (0) | 0 (0)
Solemnence (General disorders) | 0 (0) | 1 (1) | NA | 0 (0) | 0 (0) | 0 (0)
Sedation (General disorders) | 2 (2) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0)
Hypotension (General disorders) | 0 (0) | 0 (0) | NA | 1 (1) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2) | NA | 0 (0) | 0 (0) | 0 (0)
Drowsniess (General disorders) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 2 (2) | 1 (1) | NA | 2 (2) | 0 (0) | 0 (0)
Anxiety (General disorders) | 0 (0) | 1 (1) | NA | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02067975/Prot_SAP_000.pdf